CLINICAL TRIAL: NCT01177540
Title: A Randomized, Open Label, Multicenter Study to Evaluate the Efficacy and Safety of Decitabine as Epigenetic Priming With Induction Chemotherapy in Pediatric Acute Myelogenous Leukemia (AML) Subjects
Brief Title: Efficacy and Safety of Decitabine as Epigenetic Priming With Induction Chemotherapy in Pediatric Acute Myelogenous Leukemia (AML) Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to enrollment difficulties and the futility of observing differences in remission rate between treatment arms.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7373-G000-202
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2013-10

CONDITIONS: Pediatric Acute Myelogenous Leukemia (AML)
MeSH Terms: interventions — Decitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Decitabine
- Arm B (Experimental)
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 5 day priming with decitabine followed by Induction Chemotherapy of ADE (daunorubicin, cytarabine, etoposide).
  Arms: Arm A
Drug: Decitabine — Induction Chemotherapy of ADE (daunorubicin, cytarabine, etoposide) only
  Arms: Arm B

SUMMARY:
The purpose of this study is to provide data on the activity of a standard daunorubicin, cytarabine, and etoposide (ADE) induction plus epigenetic priming with decitabine as assessed by standard measures of complete remission (CR), leukemia free survival (LFS) and overall survival (OS), as well as, on minimal residual disease (MRD). It will also provide necessary data on the safety and Pharmacokinetics (PK) of decitabine in pediatric patients that is currently unavailable.

ELIGIBILITY:
Inclusion Criteria

1. Males and females, age 1 to 16 years, inclusive
2. Females of childbearing potential must have a negative serum beta human chorionic gonadotropin ( B-hCG) at Visit 1 (Screening) and a negative urine pregnancy test prior to starting study drugs (Visit 2). Female subjects of childbearing potential must agree to be abstinent or to use a highly effective method of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, intrauterine devise (IUD), or have a vasectomised partner) for at least one menstrual cycle prior to starting study drug(s) and throughout the Randomization Phase or 30 days after the last dose of study drug. Those females using hormonal contraceptives must also be using an additional approved method of contraception (as described previously)
3. Sexually mature male patients who are not abstinent or have not undergone a successful vasectomy, who are partners of women of childbearing potential must use, or their partners must use a highly effective method of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, IUD) starting for at least one menstrual cycle prior to starting study drug(s) and throughout the Randomization Phase and for 30 days (longer if appropriate) after the last dose of study drug. Those with partners using hormonal contraceptives must also be using an additional approved method of contraception (as described previously)
4. Diagnosis of acute myelogenous leukemia ( AML) (bone marrow or peripheral blood blasts greater than or equal to 20%)
5. Adequate cardiac function as defined by an echocardiogram or multiple gated acquisition (MUGA) scan demonstrating an ejection fraction greater than 50%
6. Are willing and able to comply with all aspects of the protocol
7. Provide written informed consent from subject's guardian or legally authorized representative and child assent (if applicable).

Exclusion Criteria

1. Females who are pregnant (positive B-hCG test) or lactating
2. History of chronic myelogenous leukemia (CML) [t(9;22)]
3. Acute promyelocytic leukemia (M3 subtype in French-American-British [FAB] classification)
4. Known central nervous system (CNS) leukemia
5. AML associated with congenital syndromes such as Down syndrome, Fanconi anemia, Bloom syndrome, Kostmann syndrome, or Diamond-Blackfan anemia
6. White blood cell (WBC) count greater than 100,000/mm3
7. Serum creatinine greater than 2.5 mg/dL
8. Alanine aminotransferase (ALT) greater than 5 x upper limit of normal (ULN) and/or total bilirubin greater than 3 x ULN
9. Prior chemotherapy (other than hydroxyurea) or radiation therapy for AML
10. Known to be human immunodeficiency virus (HIV) positive
11. Any history of or concomitant medical condition that, in the opinion of the Investigator, would compromise the subject's ability to safely complete the study
12. The Investigator believes the subject to be medically unfit to receive the study drug or unsuitable for any other reason
13. Subject with hypersensitivity to decitabine, daunorubicin, cytarabine, or etoposide
14. Has participated in a drug trial in the last 4 weeks.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2013-07-19 (Actual); Study Completion 2013-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Inc.
Locations (22):
- United States (17):
  - Phoenix, Arizona
  - Madera, California
  - Aurora, Colorado
  - Miami, Florida
  - Atlanta, Georgia
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Rochester, Minnesota
  - New Hyde Park, New York
  - New York, New York
  - Charlotte, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - Dallas, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- Australia (4):
  - New Lambton Heights, New South Wales
  - Westmead, New South Wales
  - Parkville, Victoria
  - Subiaco, Western Australia
- Calgary, Alberta, Canada

REFERENCES:
- [Derived] Gore L, Triche TJ Jr, Farrar JE, Wai D, Legendre C, Gooden GC, Liang WS, Carpten J, Lee D, Alvaro F, Macy ME, Arndt C, Barnette P, Cooper T, Martin L, Narendran A, Pollard J, Meshinchi S, Boklan J, Arceci RJ, Salhia B. A multicenter, randomized study of decitabine as epigenetic priming with induction chemotherapy in children with AML. Clin Epigenetics. 2017 Oct 5;9:108. doi: 10.1186/s13148-017-0411-x. eCollection 2017. PMID 29034009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 11 investigative sites in Australia, Canada and the United States from 3 March 2011 to 19 July 2013.
Pre-assignment Details: A total of 98 participants were screened, of which 25 were enrolled and treated in the study.
Groups:
- Treatment A: Decitabine + Induction Chemotherapy: Participants received decitabine 20 milligram per square meter (mg/m^2) infusion, intravenously, daily from Days 1 to 5, followed by induction chemotherapy of daunorubicin, cytarabine, etoposide for 10 days.
- Treatment B: Induction Chemotherapy Only: Participants received induction chemotherapy of daunorubicin, cytarabine, etoposide only for 10 days.
Period: Overall Study
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only
Started | 11 | 14
Completed | 10 | 14
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received at least one dose of study treatment and who had at least one postdose efficacy measurement for response.
Groups:
- Treatment A: Decitabine + Induction Chemotherapy: Participants received decitabine 20 mg/m^2 infusion, intravenously, daily from Days 1 to 5, followed by induction chemotherapy of daunorubicin, cytarabine, etoposide for 10 days.
- Total: Total of all reporting groups
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Customized [Number; unit: participants]
  1 to less than (<) 2 years | 0 | 1 | 1
  2 to 11 years | 7 | 8 | 15
  12 to 16 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 12 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Morphologic Complete Remission (CR)
Description: Disease response measurements were based on bone marrow evaluations (biopsies, aspirates, or both) performed by local pathology laboratories and assessed by study investigators. A designation of CR required that the participant achieve a morphologic leukemia-free state and have an absolute neutrophil count (ANC) greater than 1000 per microliter (/mcL) and a platelet count greater than 100,000/mcL.
Time Frame: Day 50
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only
Number analyzed (Participants) | 11 | 14
percentage of participants | 27.3 [6.0 to 61.0] | 50.0 [23.0 to 77.0]

2. Secondary Outcome: DNA Methylation
Description: Bone marrow samples were obtained at baseline and completion of induction therapy. DNA was extracted, and global DNA methylation was evaluated using the Infinium® Human Methylation450® BeadChip Array according to the manufacturer's protocol (Illumina, San Diego, California). Paired differential methylation analysis of end-induction marrows to participant matched screening marrows was performed to identify differentially methylated cytosines followed by guanine residue (CpG) loci (DML). A paired Wilcoxon rank test was conducted to compare end-induction marrows with diagnostic marrows within each arm to identify loci considered statistically significant and differentially methylated. Three different behaviors were defined: 'hypermethylation' (increased intensity in the tumor), 'hypomethylation' (decreased intensity in the tumor) and 'no change' (no substantial differences of intensity).
Time Frame: Baseline up to completion of induction therapy (Day 15)
Population: as for baseline characteristics
Measure: Count of Units; unit: Loci
Units Other Than Participants: Loci
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only
Number analyzed (Participants) | 11 | 14
Number analyzed (Loci) | 6990 | 1090
Loci
  Hypomethylated DML | 4134 | 785
  Hypermethylated DML | 2856 | 305

3. Secondary Outcome: Leukemia-free Survival (LFS)
Description: LFS was defined as time from CR until the recurrence of leukemia (greater than or equal to [>=] 5% bone marrow blasts, reappearance of peripheral blasts or the appearance of new dysplastic changes, or death, whichever occurred first). For participants who did not achieve a CR, LFS is set to zero days. For participants with CR who do not have leukemic recurrence or death, data for LFS was censored on the date of the last follow-up bone marrow or hematology examination, whichever is later. LFS was analyzed using Kaplan-Meier method.
Time Frame: Baseline to recurrence of Leukemia or Death (up to 2 years 5 months)
Population: The per protocol set included all participants who sufficiently complied with protocol. Here "overall number of participants analyzed" are participants who achieved morphologic CR and were available for this outcome measure assessment at given time period.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only
Number analyzed (Participants) | 3 | 7
days | NA [NA to NA] — There were insufficient data as of the clinical cut date to calculate median and full range from the Kaplan-Meier analysis of LFS. | NA [NA to NA] — There were insufficient data as of the clinical cut date to calculate median and full range from the Kaplan-Meier analysis of LFS.

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of study treatment to the date of death from any cause. OS was analyzed using Kaplan-Meier method.
Time Frame: Baseline to Date of Death (up to 2 years 5 months)
Population: The per protocol set included all participants who sufficiently complied with protocol.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only
Number analyzed (Participants) | 11 | 14
months | NA [6.7 to 24.5] — The median OS was not yet reached for either Treatment A or Treatment B arm at final data cutoff date. | NA [6.2 to 26.2] — The median OS was not yet reached for either Treatment A or Treatment B arm at final data cutoff date.

5. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) at Baseline and Day 50
Description: After induction chemotherapy, based on bone marrow biopsies. No formal statistical analyses of MRD were performed for this study.
Time Frame: Baseline and Day 50
Population: The full analysis set included all participants who received at least one dose of study treatment and who had at least one postdose efficacy measurement for response. Here "overall number of participants analyzed" are participants who were available for this outcome measure assessment at given time points.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only
Number analyzed (Participants) | 8 | 9
percentage of participants
  At Baseline | 75 | NA — Data was not collected and analyzed as the samples were not processed for all 9 participants due to lack of viability, degradation, or was outside established time frame for processing.
  At Day 50 | 25 | 11

6. Secondary Outcome: Time to CR
Description: Disease response measurements were based on bone marrow evaluations (biopsies, aspirates, or both) performed by local pathology laboratories an assessed by study investigators. CR: requires that the participant achieved a morphologic leukemia-free state and had an ANC >1000/mcL and platelets >100,000/mcL. Hemoglobin concentration or hematocrit had no bearing on remission status, although the participant had to be independent of transfusions. Kaplan-Meier curves were used to describe time to CR.
Time Frame: Randomization to Day 50
Population: The full analysis set included all participants who received at least one dose of study treatment and who had at least one postdose efficacy measurement for response. Here "overall number of participants analyzed" are participants who achieved morphologic CR and were available for this outcome measure assessment at given time period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only
Number analyzed (Participants) | 3 | 7
days | 43.0 [35.0 to NA] — Upper limit of 95% confidence interval (CI) could not be calculated since maximum number of participants had delayed recovery in ANC counts. | 37.0 [32.0 to 40.0]

7. Secondary Outcome: Time to Neutrophil Recovery
Description: Blood sampling was used to determine recovery, and is defined as less than or equal to 1000 per cubic millimeter (/mm^3) for absolute neutrophil count (ANC). Summarized using Kaplan-Meier product limit estimators.
Time Frame: Baseline up to Day 50
Population: The full analysis set included all participants who received at least one dose of study treatment and who had at least one postdose efficacy measurement for response. Here "overall number of participants analyzed" are participants who were available for this outcome measure assessment at given time period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only
Number analyzed (Participants) | 9 | 10
days | 26.0 [13.0 to 43.0] | 18.0 [15.0 to 25.0]

8. Secondary Outcome: Time to Platelet Recovery
Description: Blood sampling was used to determine recovery and is defined as less than or equal to 100,000/mm^3 for platelet count. Summarized using Kaplan-Meier product limit estimators.
Time Frame: Baseline up to Day 38
Population: The full analysis set included all participants who received at least one dose of study treatment and who had at least one postdose efficacy measurement for response All participants in FAS had platelet recovery.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only
Number analyzed (Participants) | 11 | 14
days | 22.0 [6.0 to 26.0] | 14.5 [8.0 to 18.0]

ADVERSE EVENTS:
Time Frame: For each participant, from the time the participant signed the informed consent form until the AE resolved, or for 30 days after the participant's last study visit, whichever came first (approximately up to 2 years and 5 months)
Arm/Group | Treatment A: Decitabine + Induction Chemotherapy | Treatment B: Induction Chemotherapy Only
All-Cause Mortality (participants affected / at risk) | 3/11 | 3/14
Serious Adverse Events (participants affected / at risk) | 2/11 | 1/14
Other Adverse Events (participants affected / at risk) | 8/11 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Decitabine + Induction Chemotherapy (N=11) | Treatment B: Induction Chemotherapy Only (N=14)
Appendicitis (Infections and infestations) | 1 | 0
Large intestine perforation (Injury, poisoning and procedural complications) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Decitabine + Induction Chemotherapy (N=11) | Treatment B: Induction Chemotherapy Only (N=14)
Anaemia (Blood and lymphatic system disorders) | 6 | 4
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2
Bradycardia (Cardiac disorders) | 1 | 2
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 3 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Caecitis (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastric fistula (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0
Lip disorder (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 2 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 5
Oral pain (Gastrointestinal disorders) | 4 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 2
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 3
Asthenia (General disorders) | 2 | 0
Catheter site discharge (General disorders) | 2 | 0
Catheter site erosion (General disorders) | 1 | 0
Catheter site erythema (General disorders) | 5 | 2
Catheter site haematoma (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 2 | 0
Catheter site oedema (General disorders) | 1 | 0
Catheter site pain (General disorders) | 3 | 3
Catheter site pruritus (General disorders) | 3 | 0
Catheter site related reaction (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Generalised oedema (General disorders) | 1 | 0
Hypothermia (General disorders) | 2 | 0
Localised oedema (General disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Nodule (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 2 | 0
Puncture site pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 2
Swelling (General disorders) | 0 | 1
Thrombosis in device (General disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Granulocyte count decreased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 3
Platelet count decreased (Investigations) | 1 | 3
Weight decreased (Investigations) | 3 | 4
Weight increased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 6 | 5
Decreased appetite (Metabolism and nutrition disorders) | 6 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 4
Lethargy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Social avoidant behaviour (Psychiatric disorders) | 1 | 0
Bladder disorder (Renal and urinary disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Penis disorder (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 1
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 5 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to enrollment difficulties and the futility of observing differences in remission rate between treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No